CLINICAL TRIAL: NCT03405363
Title: Cohort Study of Cardiovascular Events in Patients With Chronic Obstructive Pulmonary Disease Initiating Olodaterol or Other Long-acting beta2-agonists
Brief Title: Cardiovascular Events in Chronic Obstructive Pulmonary Disease Patients Initiating Olodaterol or Other Long-acting beta2 Agonists
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1222.54
Record Dates: First submitted 2018-01-15; First posted 2018-01-23 (Actual); Results first posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (2):
- new users of Olodaterol: COPD patients using Olodaterol for the first time
- new users of other LABAs: COPD patients using other long-acting beta2 agonists for the first time

SUMMARY:
Examine the risk of cardiovascular events (cardiac arrhythmia or myocardial ischemia) or all-cause mortality in Chronic Obstructive Pulmonary Disease (COPD) patients who are new users of Olodaterol or other LABAs available for the treatment of COPD.

DETAILED DESCRIPTION:
Purpose:

Time Perspective:

ELIGIBILITY:
Inclusion criteria:

* COPD diagnosis
* aged 40 years or older (to minimise the likelihood of including individuals who have asthma only)
* New user of olodaterol or a new user of indacaterol, salmeterol, or formoterol (not in fixed-dose combination with an inhaled corticosteroid) and have no dispensing of any LABA in the 6 months before the index date
* at least 1 year of enrolment in the electronic database before their first LABA dispensing (defined as the index LABA)
* Complete data on sex

Exclusion criteria:

none

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients
Sampling Method: Probability Sample
Enrollment: 65406 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2020-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Aarhus Universitets hospital Skejby, Aarhus, Denmark

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This cohort study, used data from the Danish National Patient Registry (diagnoses), Danish Prescription Database (dispensings), and Danish Register of Causes of Death (cause of death information) to examine the risk of cardiovascular events in patients with chronic obstructive pulmonary disease (COPD) exposed to olodaterol compared to other long-acting beta2-agonists (LABAs) between 01 March 2014 and 31 January 2019.
Pre-assignment Details: Only subjects that met all inclusion and none of the exclusion criteria were included. The matched cohort study design and propensity score methodology were used to establish two comparable treatment cohorts, the Olodaterol cohort and the other LABA cohort.
Groups:
- Olodaterol: Cohort of patients with Obstructive Pulmonary Disease (COPD) derived from the Danish Patient Registry initiating olodaterol (either alone or in free- or fixed-dose combination with a Long-Acting Muscarinic Antagonist (LAMA)), with first dispensing as index date occurred from 01 March 2014 (launch of olodaterol in Denmark) to 31 January 2019 (last date with data available for the final data cut).
  Participants were matched 1:4 ('olodaterol' : 'other LABAs') by age, sex, and calendar year.
- Other Long-acting beta2-agonist (LABAs): Cohort of patients with Obstructive Pulmonary Disease (COPD) derived from the Danish Patient Registry (March 2014 to January 2019) initiating LABA (alone or in a free- or fixed-dose combination with a LAMA), with first dispensing as index date occurred from 01 March 2014 (launch of olodaterol in Denmark) to 31 January 2019 (last date with data available for the final data cut).
  Participants were matched 1:4 ('olodaterol' : 'other LABAs') by age, sex, and calendar year.
Period: Overall Study
Arm/Group | Olodaterol | Other Long-acting beta2-agonist (LABAs)
Started | 14239 | 51167
Completed | 14239 | 51167
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Propensity score-trimmed population of patients with Chronic Obstructive Pulmonary Disease (COPD) derived from the Danish Patient Registry initiating olodaterol (either alone or in free- or fixed-dose combination with a LAMA) or an alternative LABA (alone or in a free- or fixed-dose combination with a LAMA).
Groups:
- Total: Total of all reporting groups
Arm/Group | Olodaterol | Other Long-acting beta2-agonist (LABAs) | Total
Number analyzed (Participants) | 14239 | 51167 | 65406
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.7 (10.0) | 72.7 (10.0) | 72.7 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7649 | 27253 | 34902
  Male | 6590 | 23914 | 30504
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of First Hospitalisation or Hospital Outpatient Clinic Visit for Atrial Fibrillation or Flutter (AF)
Description: Cases of AF were ascertained by at least one (=first occurrence) International Statistical Classification of Diseases and Related Health Problems, 10th Revision (ICD-10) code for primary hospital inpatient discharge diagnosis or as a diagnosis code in a hospital outpatient specialist visit in the Danish National Patient Registry while being new users of olodaterol or of any Long-Acting Beta2-Agonist (LABA) other than olodaterol.
  The exposure window considered only the first episode of continuous use, defined as the time comprising consecutive dispensing's separated by up to 14 days. Termination dates of the follow up: date of outcome of interest, disenrollment from the database, 14 days after estimated discontinuation of the last dispensing for index LABA, the date the patient switched to another LABA, dispensing of a second LABA, death, end of study period (= 31 January 2019).
Time Frame: Up to 4 years and 11 months
Population: Propensity score-trimmed population of patients with Chronic Obstructive Pulmonary Disease (COPD) derived from the Danish Patient Registry
Measure: Number; unit: Events
Arm/Group | Olodaterol | Other Long-acting beta2-agonist (LABAs)
Number analyzed (Participants) | 14239 | 51167
Events | 246 | 725
Statistical Analysis 1: Comparison: Olodaterol vs Other Long-acting beta2-agonist (LABAs); Test type: Other — No formal hypotheses were tested; Poisson regression model; Including exposure, natural logarithm of person-years at risk as offset, propensity score quintiles, and LAMA use at the index date as a covariate; Adjusted Incidence Rate Ratio = 1.20, 95% CI 2-sided [0.98 to 1.47] — Olodaterol compared to 'other LABA' as reference

2. Primary Outcome: Occurrence of First Hospitalisation or Hospital Outpatient Clinic Visit for Supraventricular Tachycardia (SVT) (Other Than Atrial Fibrillation/Flutter)
Description: Cases of SVT were ascertained by at least one (=first occurrence) ICD-10 code for primary hospital inpatient discharge diagnosis or as a diagnosis code in a hospital outpatient specialist visit in the Danish National Patient Registry while being new users of olodaterol or of any Long-Acting Beta2-Agonist (LABA) other than olodaterol.
  The exposure window considered only the first episode of continuous use, defined as the time comprising consecutive dispensing's separated by up to 14 days. Termination dates of the follow up: date of outcome of interest, disenrollment from the database, 14 days after estimated discontinuation of the last dispensing for index LABA, the date the patient switched to another LABA, dispensing of a second LABA, death, end of study period (= 31 January 2019).
Time Frame: Up to 4 years and 11 months
Population: as for outcome 1
Measure: Number; unit: Events
Arm/Group | Olodaterol | Other Long-acting beta2-agonist (LABAs)
Number analyzed (Participants) | 14239 | 51167
Events | 19 | 38
Statistical Analysis 1: Comparison: Olodaterol vs Other Long-acting beta2-agonist (LABAs); No formal hypotheses were tested; Test type: Other; Poisson regression model; [statistical method as in outcome 1, analysis 1]; Adjusted Incidence Rate Ratio = 1.83, 95% CI 2-sided [0.90 to 3.74] — Olodaterol compared to 'other LABA' as reference

3. Primary Outcome: Occurrence of First Hospitalisation for Ventricular Tachycardia (VT), Including Ventricular Fibrillation/Flutter and Cardiac Arrest
Description: Cases of VT were ascertained by at least one (=first occurrence) ICD-10 code for primary hospital inpatient discharge diagnosis in the Danish National Patient Registry while being exposed to olodaterol and other LABA monotherapy or in free or fixed-dose combination with long-acting muscarinic antagonist (LAMA).
  The exposure window considered only the first episode of continuous use, defined as the time comprising consecutive dispensing's separated by up to 14 days. Termination dates of the follow up: date of outcome of interest, disenrollment from the database, 14 days after estimated discontinuation of the last dispensing for index LABA, the date the patient switched to another LABA, dispensing of a second LABA, death, end of study period (= 31 January 2019).
Time Frame: Up to 4 years and 11 months
Population: as for outcome 1
Measure: Number; unit: Events
Arm/Group | Olodaterol | Other Long-acting beta2-agonist (LABAs)
Number analyzed (Participants) | 14239 | 51167
Events | 29 | 80
Statistical Analysis 1: Comparison: Olodaterol vs Other Long-acting beta2-agonist (LABAs); No formal hypotheses were tested; Test type: Other; Poisson regression model; [statistical method as in outcome 1, analysis 1]; Adjusted Incidence Rate Ratio = 1.30, 95% CI 2-sided [0.71 to 2.36] — Olodaterol compared to 'other LABA' as reference

4. Primary Outcome: Occurrence of First Hospitalisation for Acute Myocardial Infarction (AMI)
Description: Cases of AMI were ascertained by at least one (=first occurrence) ICD-10 code for primary hospital inpatient discharge diagnosis in the Danish National Patient Registry while being new users of olodaterol or of any Long-Acting Beta2-Agonist (LABA) other than olodaterol.
  The exposure window considered only the first episode of continuous use, defined as the time comprising consecutive dispensing's separated by up to 14 days. Termination dates of the follow up: date of outcome of interest, disenrollment from the database, 14 days after estimated discontinuation of the last dispensing for index LABA, the date the patient switched to another LABA, dispensing of a second LABA, death, end of study period (= 31 January 2019).
Time Frame: Up to 4 years and 11 months
Population: as for outcome 1
Measure: Number; unit: Events
Arm/Group | Olodaterol | Other Long-acting beta2-agonist (LABAs)
Number analyzed (Participants) | 14239 | 51167
Events | 56 | 137
Statistical Analysis 1: Comparison: Olodaterol vs Other Long-acting beta2-agonist (LABAs); No formal hypotheses were tested; Test type: Other; Poisson regression model; [statistical method as in outcome 1, analysis 1]; Adjusted Incidence Rate Ratio = 1.22, 95% CI 2-sided [0.79 to 1.87] — Olodaterol compared to 'other LABA' as reference

5. Primary Outcome: Occurrence of First Hospitalisation for Serious Acute Coronary Heart Disease (SACHD), Including Angina and Other Acute Ischaemic Heart Disease Events
Description: Cases of SACHD were ascertained by at least one (=first occurrence) ICD-10 code for primary hospital inpatient discharge diagnosis in the Danish National Patient Registry while being new users of olodaterol or of any Long-Acting Beta2-Agonist (LABA) other than olodaterol.
  The exposure window considered only the first episode of continuous use, defined as the time comprising consecutive dispensing's separated by up to 14 days. Termination dates of the follow up: date of outcome of interest, disenrollment from the database, 14 days after estimated discontinuation of the last dispensing for index LABA, the date the patient switched to another LABA, dispensing of a second LABA, death, end of study period (= 31 January 2019).
Time Frame: Up to 4 years and 11 months.
Population: as for outcome 1
Measure: Number; unit: Events
Arm/Group | Olodaterol | Other Long-acting beta2-agonist (LABAs)
Number analyzed (Participants) | 14239 | 51167
Events | 41 | 147
Statistical Analysis 1: Comparison: Olodaterol vs Other Long-acting beta2-agonist (LABAs); No formal hypotheses were tested; Test type: Other; Poisson regression model; [statistical method as in outcome 1, analysis 1]; Adjusted Incidence Rate Ratio = 1.00, 95% CI 2-sided [0.64 to 1.56] — Olodaterol compared to 'other LABA' as reference

6. Secondary Outcome: All-cause Mortality.
Description: Death ascertained from Danish Civil Registration System (fact and date of death, but not cause of death) while being new users of olodaterol or any Long-Acting Beta2-Agonist (LABA) other than olodaterol.
  Exposure window: first episode of continuous use (= time comprising consecutive dispensing's separated by up to 14 days). Termination dates of the follow up: date of outcome of interest, disenrollment from database, 14 days after estimated discontinuation of last dispensing for index LABA, date patient switched to another LABA, dispensing of a second LABA, death, end of study period (= 31 January 2019).
  To assess possible impact of imbalanced baseline characteristics, all-cause mortality was further assessed in two post-hoc analyses with restricted populations that would be more similar at baseline, post-hoc population 1 and post-hoc population 2.
Time Frame: Up to 4 years and 11 months.
Population: Propensity score-trimmed population of patients with Chronic Obstructive Pulmonary Disease (COPD) derived from the Danish Patient Registry. Post-hoc population 1 was based on propensity score-trimmed population restricted to users of fixed-dose combination of LABA/LAMA who were LABA-treatment naïve (= no LABA dispensing in the 180 days before cohort entry). Post-hoc population 2 was post-hoc population 1 further restricted to users without hospitalizations for COPD in the last 90 days.
Measure: Number; unit: Events
Arm/Group | Olodaterol | Other Long-acting beta2-agonist (LABAs)
Number analyzed (Participants) | 14239 | 51167
Events | 859 | 1872
Statistical Analysis 1: Comparison: Olodaterol vs Other Long-acting beta2-agonist (LABAs); Analysis was based on Propensity score-trimmed population of patients with Chronic Obstructive Pulmonary Disease (COPD) derived from the Danish Patient Registry; Test type: Other — No formal hypotheses were tested; Poisson regression model; [statistical method as in outcome 1, analysis 1]; Adjusted Incidence Rate Ratio = 1.63, 95% CI 2-sided [1.44 to 1.84] — Olodaterol compared to 'other LABA' as reference
Statistical Analysis 2: Comparison: Olodaterol vs Other Long-acting beta2-agonist (LABAs); Analysis based on post-hoc population 1. Adjustments: propensity score decile, previous use of: LAMA, oxygen, inhaled glucocorticoid, respiratory medications, fixed-dose combinations of Short-Acting Beta2- Agonist and Short-Acting Muscarinic Antagonist and systemic antibacterials. COPD severity, number of: all-cause hospitalisations 365 and 180 days, COPD exacerbations 180 and 90 days, COPD hospitalisations 180 and 90 days, and COPD exacerbations 90 days before index date; Test type: Other — No formal hypotheses were tested; Poisson regression model; Adjusted Incidence Rate Ratio = 1.48, 95% CI 2-sided [1.23 to 1.78] — Olodaterol compared to 'other LABA' as reference
Statistical Analysis 3: Comparison: Olodaterol vs Other Long-acting beta2-agonist (LABAs); Analysis based on post-hoc population 2. Adjustments: propensity score decile, previous use of: LAMA, oxygen, inhaled glucocorticoid, respiratory medications. COPD severity, number of all-cause hospitalisations 180 days, COPD exacerbations 180 days before cohort entry; Test type: Other — No formal hypotheses were tested; Poisson regression model; Adjusted Incidende Rate Ratio = 1.26, 95% CI 2-sided [0.97 to 1.64] — Olodaterol compared to 'other LABA' as reference

ADVERSE EVENTS:
Time Frame: Up to 4 years and 11 months
Description: This is a non-interventional study using electronic health care records, with data retrieved from Danish National Patient Registry, Danish National Prescription Registry and Danish Register of Causes of Death. No adverse events were collected on an individual case level.
  All-cause mortality (ACM) is an outcome of this study and thus additionally reported below. Please note, adjusted incidence rate ratios of ACM are displayed as statistical analyses 1, 2, 3 of the secondary outcome measure 6.
Arm/Group | Olodaterol | Other Long-acting beta2-agonist (LABAs)
All-Cause Mortality (participants affected / at risk) | 859/14239 | 1872/51167
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-28): https://cdn.clinicaltrials.gov/large-docs/63/NCT03405363/Prot_SAP_000.pdf